CLINICAL TRIAL: NCT03479151
Title: Magnetic Resonance Guided High Intensity Focused Ultrasound (MRgHIFU) for Pain Palliation of Bone Metastases
Acronym: HIFU-Bone
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: CI of study retired on 6.10.2020 and there will be no further efforts to apply for an extension in order to recruit to this study.
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Philips Medical Systems (Industry); Cancer Research UK (Other)
Responsible Party: Principal Investigator, Nandita deSouza, Professor Nandita Da Souza, Institute of Cancer Research, United Kingdom
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17/LO/1689 CCR 4733
Record Dates: First submitted 2018-02-27; First posted 2018-03-27 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Cancer; Bone Metastases
Keywords: Magnetic Resonance Imaging (MRI); High Intensity Focused Ultrasound (HIFU)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-HIFU of painful bone metastases (Experimental): Magnetic Resonance guided High Intensity Focused Ultrasound (MRgHIFU) for Pain Palliation of Bone Metastases
  Interventions: Device: Magnetic Resonance Image-guided High Intensity Focused Ultrasound (MR-HIFU)

INTERVENTIONS:
Device: Magnetic Resonance Image-guided High Intensity Focused Ultrasound (MR-HIFU) — MRgHIFU treatment will be delivered using a Philips Sonalleve system, which integrates a high intensity phased array focused ultrasound transducer with our Philips 3T Achieva imaging system. An electromechanical transducer positioning system is used to deliver spatially and temporally controlled ultrasound energy and thermal heat to tissues non-invasively. The MR system is used to provide images to plan the therapy, and to guide and monitor the thermal ablation with thermal imaging during the treatment.

SUMMARY:
The primary objective of this study is to determine whether intra- and post-procedural MR changes are indicative of reduction in pain symptom scores. The trial will recruit a cohort of patients with painful bone metastases, who wish to consider MRgHIFU treatment. These patients will be identified in conjunction with the pain and palliative care teams, as well as clinical and medical oncologists. Patients will undergo MRgHIFU treatment using scanning and treatment planning methods that have been established in the patients treated within the multi-centre study. The treatment response rate for the cohort will be recorded. Intra- and post-procedural imaging metrics will be evaluated for their ability to detect tissue changes, which may be indicative of response. Patients will be followed-up for up to 90 days after treatment, and will attend for repeat imaging and pain review at days 30, 60 and 90 after treatment. Any changes in imaging metrics will be compared between responders and non-responders.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate whether the ablated tissue volume indicated by immediate post-treatment Gd-T1W imaging is indicative of reduction in pain scores (response) 30 days after treatment.

The secondary aims of this study are:

* To record the proportion of patients responding to MRgHIFU treatment at Days 7, 14, 30, 60 and 90 after treatment
* To investigate whether intra-procedural PRFS metrics (thermal dose volume, temperature) are indicative of subsequent treatment response
* To investigate whether intra- or post-procedural changes in ADC or T2 are indicative of subsequent treatment response
* To record adverse events arising as a result of MRgHIFU treatment
* To evaluate the effect of MRgHIFU treatment on patients' quality of life
* To record the time to pain progression and the duration of pain response for patients in this cohort
* To estimate the costs of MRgHIFU treatment

This is an exploratory study, which will recruit n=15 patients into one single cohort. Enrolment of the target population for the study is expected to take approximately 2 years. Patients will be eligible for the study if they wish to consider MRgHIFU treatment for pain palliation of a region of bony metastatic disease that is accessible to the MRgHIFU device. After providing their written informed consent to participate in the study, patients' suitability for treatment will be determined by a combined assessment of clinical review by a pain specialist, and an MR screening investigation to establish lesion targetability. Baseline clinical and imaging metrics will be recorded. Patients who fulfill all inclusion criteria, have none of the exclusion criteria, and who give informed consent, will be scheduled for MRgHIFU treatment to the target lesion. Treatment will be delivered under sedation on a day-case basis, according to protocols already established in our prior study. During treatment delivery, the investigators will assess imaging metrics of tissue change, which may be indicative of subsequent treatment response. Treatment would be expected to take approximately 1-2 hours, and after an observation period of approximately 2-4 hours, the patient will be discharged. Before discharge, follow-up instructions will be given to the patient. Patients' clinical and imaging responses to treatment will then be assessed at follow-up appointments up to 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful bony metastatic disease
* Target bony metastatic lesion is painful (NRS≥4)
* Intended target region accessible for MRgHIFU treatment (usually not skull or spinal metastases above the sacrum)
* Intended target region visible on non-contrast MR imaging

Exclusion Criteria:

* MRI contra-indicated (e.g. by incompatible metal implants, claustrophobia, or because BMI precludes accommodation in the MR scanner)
* Pregnancy
* Sedation contra-indicated
* Critical anatomical structure cannot be avoided along the beam path or the at the target (can be assessed at screening)
* Internal or external fixation device along the beam path or at the target

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Measure the ablated tissue volume indicated by immediate post-treatment Gd-T1W imaging in responders and non-responders. | Day 30

SECONDARY OUTCOMES:
To report the treatment response rate. | up to 90 days
  Days 7, 14, 30, 60 and 90
To investigate whether ablated tissue volume indicated by Gd-T1W imaging at Day 30 remains stable at Days 60 and 90. | up to 90 days
.To investigate whether intra-procedural PRFS metrics are different in responders and non-responders at Day 30 | 30 days post treatment
  PRFS Metrics include thermal dose volume, temperature
To investigate whether intra- or post-procedural changes in ADC are different in responders and non-responders. | Day 30
To investigate whether intra- or post-procedural changes in T2 are different in responders and non-responders. | Day 30
The rate of treatment-related adverse events | up to 3 months after treatment.
The effect of MRgHIFU treatment on patients' quality of life, recorded using Quality of Life Questionnaires (QLQ's). | up to 3 months after treatment.
  using EORTC (European Organization for Research and Treatment of Cancer)- QLQ's
The costs of MRgHIFU treatment. | up to 3 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nandita deSouza, Professor, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom